CLINICAL TRIAL: NCT00162214
Title: Phase I Study to Evaluate the Effect of Ketoconazole on the Pharmacokinetics of Dasatinib and the Effect of Dasatinib on Pharmacodynamic Markers in Patients With Advanced Solid Tumors
Brief Title: Study of Dasatinib in Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA180-021
Record Dates: First submitted 2005-09-09; First posted 2005-09-13 (Estimated); Last update posted 2011-04-14 (Estimated); Status verified 2011-04

CONDITIONS: Tumors
Keywords: Advanced Solid Tumors
MeSH Terms: conditions — Neoplasms | interventions — Dasatinib; Ketoconazole

ARMS (1):
- 1 (Active Comparator)
  Interventions: Drug: Dasatinib + Ketoconazole

INTERVENTIONS:
Drug: Dasatinib + Ketoconazole — Tablets, Oral, Segment 1: escalating single dose of dasatinib starting at 140 mg q24 hours on Day 1-8; single dose of ketoconazole 200 mg q12 hours on Days 3-8; Segment 2: single daily oral doses of dasatinib, once daily, until disease progression or unacceptable toxicity.
  Other Names: Sprycel

SUMMARY:
The purpose of Segment 1 of the study is to determine the effect of ketoconazole on dasatinib. The purpose of Segment 2 is to learn how dasatinib affects tumor growth in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* ECOG status 0-2
* Advanced or metastatic disease, unresponsive to standard treatment (or no standard treatment exists)
* Biopsy pretreatment
* Adequate bone marrow, liver and kidney function

Exclusion Criteria:

* Serious cardiovascular disease
* Bleeding disorders
* Gastrointestinal (GI) tract disease
* Platelet inhibitors
* H2 blockers, proton pump inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2005-08; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Segment 1: Determine whether the steady state pharmacokinetics of 20 mg of dasatinib are affected by co-administration with ketoconazole in patients with advanced solid tumors
Segment 2: Assess the pharmacodynamic activity of dasatinib

SECONDARY OUTCOMES:
Segment 1: Evaluate the safety and tolerability of dasatinib alone and when co-administered with ketoconazole
Segment 2: Explore the association between tumor response and the pre-clinically identified markers and other mRNA gene expression level

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Lee S. Rosen M.D., Santa Monica, California
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Md Anderson Cancer Center, Houston, Texas